CLINICAL TRIAL: NCT03666221
Title: An Open,Multicenter,Phase II Trial of Intensity Modulated Radiation Therapy Combined With Concurrent Nimotuzumab in Patient With Recurrent Nasopharyngeal Carcinoma
Brief Title: Nimotuzumab for Recurrent Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Sun Yat-sen University (Other); Jiangxi Provincial Cancer Hospital (Other); Zhejiang Cancer Hospital (Other); Fujian Medical University Union Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC001.2
Record Dates: First submitted 2018-09-10; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Recurrent Nasopharyngeal Carcinoma
Keywords: Nimotuzumab; IMRT; Radiation; Recurrent; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence | interventions — nimotuzumab; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nimotuzumab plus IMRT (Experimental): Patients with recurrent nasopharyngeal carcinoma were given an initial dose of nimotuzumab (200 mg) 7days before receiving concurrent intensity modulated radiation therapy(IMRT) , folowing weekly nimotuzumab (200 mg/week) for totally 8 weeks concurrent with IMRT.
  Interventions: Drug: Nimotuzumab

INTERVENTIONS:
Drug: Nimotuzumab — Drug: Nimotuzumab Radiation: Intensity Modulated Radiation Therapy
  Other Names: Radiation

SUMMARY:
The study assessed the clinical efficacy, and safety of the combination of Nimotuzumab administered concomitantly with intensity modulated radiation therapy(IMRT) in patients with recurrent nasopharyngeal cancer.

DETAILED DESCRIPTION:
The clinical efficacy of Nimotuzumab combined with radiotherapy has been shown in advanced nasopharyngeal cancer, which was significantly higher than radiotherapy alone. The efficacy of radiotherapy combined with Nimotuzumab has not been confirmed in recurrent nasopharyngeal cancer.In this study, Phase II clinical trials were performed. The patients were treated with Nimotuzumab which were used concurrently with IMRT. The efficacy and toxicity will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent tumor in nasopharynx with or without relapse cervical lymph nodes more than 6 months after initial radical treatment.
2. Recurrent nasopharyngeal cancer was confirmed by pathology, marginal recurrence can be diagnosed by imaging examinations.
3. Age 18-70.
4. At least one of the tumor lesions measurable.
5. Functional Status: PS (ECOG) > 0-1.
6. Normal Bone Marrow Function: White blood cell count > 4×109/L, hemoglobin >90g/L, and platelet count >100×109/L.
7. Normal Hepatic and Renal Function: Alanine Tminotransferase (ALT)/Aspartate Aminotransferase (AST) < 2.5 times the upper limit of normal (ULN), while total bilirubin (T-Bil) < 1.5 x ULN and serum creatinine < 1.5 x ULN.
8. Life expectancy of more than 6 months.
9. All the patients signed the informed consent.
10. Follow up regularly and comply with test requirements.

Exclusion Criteria:

1. Patients with recurrent cervical lymph nodes alone.
2. Evidence of distant metastasis
3. The relapse tumor has been treated with chemotherapy, radiotherapy, surgery, immunotherapy and other anti-tumor therapy.
4. Creatinine clearance < 30ml/min
5. Has received epidermal growth factor targeting therapy.
6. Second malignancy within 5 years(except of Non-melanoma Skin Cancer or carcinoma in situ of cervix).
7. Serious complications, such as uncontrolled hypertension, coronary heart disease, diabetes, heart failure, etc.
8. Active systemic infection.
9. History of Serious lung or heart disease.
10. Drug or alcohol addiction.
11. Persons without capacity for civil conduct or persons with limited capacity for civil conduct.
12. The patient has physical or mental disorders and is believed to be unable to fully or fully understand the possible complications of the study.
13. To receive chronic systemic immunotherapy or hormone therapy other than this study.
14. Women who are pregnant or breast feeding
15. Participation in other drugs clinical trials within 1 month.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2014-11-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Tumor response rate after Nimotuzumab concurrent with radiotherapy for recurrent NPC patients | Three month after patients subject to the treatment
  The response status (Complete Response + Partial Response) was evaluated according to RECIST (Response Evaluation Criteria in Solid Tumors) criteria. Complete response was defined as disappearance of all target lesions, and Partial response was defined as at least a 30% reduction in the sum of the longest diameter of target lesions, taking as reference the baseline study.
Toxicity of this combined treatment for recurrent NPC patients | Three month after patients subject to the treatment
  Adverse events of this combined modality treatment were graded according to CTCAE (Common Terminology Criteria for Adverse Events) v3.0 criteria.Toxicity Criteria for Adverse Events version 3.0

SECONDARY OUTCOMES:
Local Progression free survival | Three years
Disease-free survival | Three years
  Defined as the time in month from all treatment were finished to the date of disease progress is observed.
Overall survival | Three years
  Defined as the time in month from diagnosis of recurrent NPC to the date of death is observed or to last follow-up visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of radiation oncology, Fujian cancer hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No